CLINICAL TRIAL: NCT02051426
Title: Behavioral and Cognitive Effects of the N-methyl-D-aspartate Receptor (NMDAR) Co-agonist D-serine in Healthy Humans
Acronym: NMDAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herzog Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 112-06
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: neuropsychiatric effects
MeSH Terms: interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-serine (Experimental): single P.O. administration of D-serine (2.1g)
  Interventions: Other: D-serine
- Placebo (Placebo Comparator): single P.O. administration of corn starch
  Interventions: Other: Placebo

INTERVENTIONS:
Other: D-serine — single P.O. administration of D-serine (2.1g)
  Other Names: DSR
  Arms: D-serine
Other: Placebo — single P.O. administration of Placebo
  Other Names: corn starch
  Arms: Placebo

SUMMARY:
The efficacy of compounds having agonistic activity at the glycine site associated with the N-methyl-D-aspartate receptor (NMDAR) is presently assessed in psychiatric disorders. In contrast to NMDAR antagonists, the neuropsychiatric effects of NMDAR agonists in the healthy human organism are not known. The investigators studied neuropsychiatric and neurochemical effects of the NMDAR-glycine site obligatory co-agonist D-serine (DSR) in healthy subjects using a randomized, controlled crossover challenge design including a baseline assessment day and two treatment administration days (DSR and placebo in randomized order). Thirty-five subjects aged 23-29 years participated in the study and received a 2.1g orally administered DSR dose. The main outcome measures were the changes in scores of mood-related Visual Analogue Scale (VAS), Continuous Performance Test - Identical Pairs (CPT-IP), and Rey Auditory Verbal Learning Test (RAVLT).

DETAILED DESCRIPTION:
The study employed a randomized, double-blind, placebo controlled crossover design according to which, following a baseline assessment session, subjects were tested under two acute treatment conditions on two separate days. Following the baseline assessment day, 16 subjects were randomized, using a computer-generated random number sequence, to receive during test day 1 DSR and 19 to receive placebo. During test day 2, these two groups of subjects were crossed over to receive the alternative experimental treatment. The time intervals between the baseline assessment day, test day 1 and test day 2 were two to three weeks and 1 month respectively, in order to avoid the possibility of any carry-over effects.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* history of psychiatric, medical, neurological illness or substance abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2007-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Heresco-Levy, M.D., Principal Investigator — Herzog Hospital

REFERENCES:
- [Derived] Levin R, Dor-Abarbanel AE, Edelman S, Durrant AR, Hashimoto K, Javitt DC, Heresco-Levy U. Behavioral and cognitive effects of the N-methyl-D-aspartate receptor co-agonist D-serine in healthy humans: initial findings. J Psychiatr Res. 2015 Feb;61:188-95. doi: 10.1016/j.jpsychires.2014.12.007. Epub 2014 Dec 24. PMID 25554623

RESULTS

PARTICIPANT FLOW:
Groups:
- D-serine First, Then Placebo: D-serine (2.1g), then Placebo (corn starch)
- Placebo First, Then D-serine: corn starch, then D-serine (2.1g)
Period: First Intervention
Arm/Group | D-serine First, Then Placebo | Placebo First, Then D-serine
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0
Period: Washout Period of 1 Month
Arm/Group | D-serine First, Then Placebo | Placebo First, Then D-serine
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | D-serine First, Then Placebo | Placebo First, Then D-serine
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 16 participants received DSR then 1month later received placebo; whereas19 participants received placebo then 1 month later received DSR. The assessments were performed at baseline assessment day and 2 hours after the experimental treatment administration (test day1&2). Outcome analysis was D-serine versus Placebo effects for total 35 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | D-serine First, Then Placebo | Placebo First, Then D-serine | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.58 (3.0) | 26.58 (3.0) | 26.58 (3.0)
Sex/Gender, Customized [Number; unit: participants]
  female | 5 | 8 | 13
  male | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analogue Scale (VAS) of Anxiety - From Baseline to 2 Hours
Description: The subject was asked to point on the VAS scale according to his anxiety level. VAS anxiety scale 0 to 10 ( 0 [no anxiety] to 10 [maximum anxiety] ).
Time Frame: Baseline, 2 hours post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- D-serine: D-serine (2.1g)
- Placebo: corn starch
Arm/Group | D-serine | Placebo
Number analyzed (Participants) | 35 | 35
units on a scale | 0.5 (0.2) | 0.0 (0.2)

2. Primary Outcome: Change in Cognitive Function- CPT-IP D-prime Score - From Baseline to 2 Hours
Description: The "d-prime score" is a score given to each participant on a scale of 0.0 - 1.0 in which discrimination sensitivity is measured. A score of 0 equates to no sensitivity whereas a score of 1.0 equates to perfect sensitivity.
Time Frame: Baseline, 2 hours post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine | Placebo
Number analyzed (Participants) | 35 | 35
units on a scale | .5 (.2) | 0 (.2)

3. Primary Outcome: Change in Rey Auditory Verbal Learning Test RAVLT (Trial 7) - From Baseline to 2 Hours
Description: RAVLT measures short term verbal memory, verbal learning, susceptibility to (proactive and retroactive) interference, retention of information after a certain period of time during which other activities are performed and recognition memory. The test consists of a list of 15 common nouns, which are read to the subject in five consecutive trials (trials 1 through 5); each reading is followed by a free-recall task. In trial 6, an interface list of 15 new common nouns is presented, followed by free recall of these new nouns. In trial 7, without additional reading, subjects are again asked to recall the first list. Twenty minutes later, without an additional reading, subjects are asked to recall once more the first list (trial 8). The RAVLT score range from 0-90 correctly recalled words. For trial 7 the score ranges from 0 to 15 correctly recalled words.
Time Frame: Baseline, 2 hours post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine | Placebo
Number analyzed (Participants) | 35 | 35
units on a scale | 2 (.3) | .3 (.3)

ADVERSE EVENTS:
Time Frame: at the end of test days 1 and 2
Description: Udvalg for Kliniske Undersogelser (UKU) Side Effects Rating Scale
Arm/Group | D-serine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes